CLINICAL TRIAL: NCT07315165
Title: A Phase II Randomized Trial of Enteral Nutrition Versus Standard of Care in Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Enteral Nutrition Versus Standard of Care in Allogeneic Hematopoietic Stem Cell Transplantation
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ENABLE
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplant (Allo-HSCT)
Keywords: Enteral Nutrition; Acute GVHD; Stage 3-4; Stage 2-4 Gut GVHD; Nutritional Support; allo-HSCT.
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Intervention Model Description: All patients in both arms will receive nutrition counseling regarding the use of a high-protein, high-energy diet with snacks and high-protein supplement drinks, as tolerated.
  Two groups will be randomized, one receiving standard of care and the other receiving eteral nutrition via nasogastric tube. Outcomes will be compared between the two groups.
  In the study group, enteral nutrition will be administered, starting on allo-HSCT day +1 (the day after the infusion of stem cell transplant). Enteral nutrition will be administered through an enteral nutrition tube; the most commonly used equipment is a nasogastric tube of 8-10 Fr gauge.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control (initiation of supplemental enteral or parenteral nutrition as clinically indicated) (Active Comparator)
  Interventions: Dietary Supplement: Enteral Nutrition
- The study group (enteral nutrition starting on day +1) (Experimental)
  Interventions: Dietary Supplement: Enteral Nutrition

INTERVENTIONS:
Dietary Supplement: Enteral Nutrition — A commercially available blenderized tube feed nutrition (BTF) formula will be initiated at a fixed starting rate of 25 ml/hr. The infusion rate will be increased in consultation with a registered dietitian nutritionist (RDN) based on tolerance to reach a feeding goal of 30-35 kcal/kg/day, which includes 1.5-2 g of protein/kg/day.

SUMMARY:
This is a randomized controlled phase II trial which will enroll 112 patients with a diagnosis of a blood cancer or a serious blood disorder who plan to undergo an allogenic hematopoietic stem cell transplant using any conditioning regimen or graft source. Eligible patients will be randomized to receive standard of care (e.g., initiation of supplemental nutrition when oral intake declines) versus enteral nutrition via enteral feeding tube starting on day +1 post-transplant for at least 7 days, usually until engraftment. The primary endpoint will be cumulative incidence of stage 3-4 acute GVHD of the lower gut by day +100 post-transplant, whereas secondary endpoints will be stage 2-4 acute GVHD of the lower gut by day +100, grade 2-4 acute GVHD, weight loss and changes in lean muscle mass, changes in physical function, health-related quality of life, length of transplant hospital stay, and time to platelet and neutrophil engraftment. Assessments will include acute GVHD assessments and grading, Activities of Daily Living (ADL), Instrumental Activities of Daily Living (IADL), Fried Frailty Index, and Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a hematological condition or serious blood disorder
* Patient planned for an allogeneic hematopoietic stem cell transplant
* Any conditioning regimen or graft source

Exclusion Criteria:

* Uncorrected anatomical deformity of the nose, nasopharynx, esophagus, or stomach that could prevent proper placement of a nasogastric tube.
* Chronic gastrointestinal conditions causing malabsorption or need for nutritional supplementation, e.g., celiac disease, short gut syndrome, chronic use of total parental nutrition or enteral nutrition for 3 or more months. Uncorrected anatomical deformity may include any known significant deviated nasal septum, large nasal polyps or other masses, or nasal or oropharyngeal trauma.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Stage 3-4 Acute GVHD of Lower Gut | 100 Days post- transplant
  Cumulative incidence will be calculated as the time to stage 3-4 acute GVHD of the lower gut for each of the study arms.

SECONDARY OUTCOMES:
Incidence of Stage 2-4 Acute GVHD of Lower Gut | 100 Days post- transplant
  Cumulative incidence will be calculated as the time to stage 2-4 acute GVHD of the lower gut for each of the study arms
Percent change in weight | Day +30 and Day +100 post-transplant
  Percent change from baseline weight at day +30 and day +100 post-transplant.
Percent change in lean body mass | Baseline and Day +30 post-transplant
  Percent change in total lean body mass measured by DEXA scan at baseline and day +30 post-transplant.
Health-Related Quality of Life (HRQoL) | Baseline and Day +100 post-transplant
  Functional Assessment of Cancer Therapy - Bone Marrow Transplant (FACT-BMT), total score range 0-148, where higher scores indicate better quality of life.
Transplant hospital stay | Up to approximately 30 Days Post Transplant
  Median duration of transplant hospital stay compared between groups.
Platelet and neutrophil engraftment | Aproximately14 days post-transplant
  Cumulative incidence curves of platelet engraftment and neutrophil engraftment will be generated using the methods of Gray to adjust for the competing risk of death to determine the probabilities of neutrophil and platelet engraftment.
Functional status and physical performance | Day +30, and Day +100 post-transplant
  Fried Frailty Index score ranges from 0 to 5, where higher scores indicate greater frailty (worse functional status).
Functional status and physical performance Activities of Daily Living (ADL) | Day +30, and Day +100 post-transplant
  Change in Activities of Daily Living (ADL) score from baseline to Day +30 and Day+100 post-transplant.
  The ADL scale ranges from 0 to 6, where higher scores indicate greater independence (better functional status).
Functional status and physical performance Instrumental Activities of Daily Living (IADL) | Day +30, and Day +100 post-transplant
  Change in Instrumental Activities of Daily Living (IADL) score from baseline to Day +30 and Day +100 post - transplant.
  The IADL score ranges from 0 to 8, where higher scores indicate greater independence (better functional status).
Functional status and physical performance | Day +30, and Day +100 post-transplant
  Karnofsky Performance Scale ranges from 0 to 100, where higher scores indicate better functional status.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Haddadin, MD, Principal Investigator — University of Nebraska
Locations (1):
- Fred & Pamela Buffet Cancer Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No